CLINICAL TRIAL: NCT06183229
Title: Double-blind Placebo-controlled Randomized Trial of Efficacy and Safety of Cycloferon, Enteric-coated Tablets, 150 mg, for Post-exposure Prophylaxis of Acute Respiratory Viral Infection and Influenza
Brief Title: Cycloferon for Post-exposure Prophylaxis of Acute Respiratory Viral Infections and Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCF-III-TAB-2023
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-01

CONDITIONS: Influenza; Acute Respiratory Infection
Keywords: influenza; acute respiratory viral infection; grippe; prevention
MeSH Terms: conditions — Influenza, Human | interventions — 10-carboxymethyl-9-acridanone

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized, two-parallel group comparative study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization is performed using the Internet Interactive Response System (IWRS) before the start of the drug dosing period. During the randomization procedure, the investigator, after assessing whether the subject meets the inclusion criteria and the absence of non-inclusion criteria, will contact IWRS, the system will record the fact that the subject has been randomized and will automatically report the package number of the drug that must be given to the subject.
  The study drug CYCLOFERON®, enteric-coated tablets, 150 mg (NTFF POLYSAN LLC, Russia), is supplied in the form of enteric-coated tablets, 150 mg. 10 tablets in a blister pack, 5 blister packs in a cardboard box.
  The reference drug PLACEBO, enteric-coated tablets, 150 mg (NTFF POLYSAN LLC, Russia), is supplied in the form of enteric-coated tablets, 150 mg. 10 tablets in a blister pack, 5 blister packs in a cardboard box.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cycloferon (Experimental): Intake of Cycloferon, enteric-coated tablets, 150 mg, 4 tablets (600 mg) per day on days 1, 2, 4, 6 and 8.
  Interventions: Drug: Cycloferon
- Placebo (Placebo Comparator): Intake of Placebo, 4 tablets per day, on days 1, 2, 4, 6 and 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cycloferon — Cycloferon, enteric-coated tablets, 150 mg, 4 tablets (600 mg) per day on days 1, 2, 4, 6 and 8.
  Other Names: Meglumine acridоnacetate
  Arms: Cycloferon
Drug: Placebo — Placebo tablets, 4 tablets per day on days 1, 2, 4, 6 and 8
  Arms: Placebo

SUMMARY:
Influenza and other acute respiratory viral infections remain practically uncontrollable diseases due to the high variability of the antigenic structure of influenza viruses and the heterogeneity of pathogens of acute respiratory infections. Therefore, for the prevention and treatment of influenza, acute respiratory viral infections and herpes infections, it is relevant to develop drugs - immunomodulators that mobilize the reserves of nonspecific and specific immune systems and enhance the effects of these systems against the pathogens. The drug CYCLOFERON, 150 mg, enteric-coated tablets, contains the active substance meglumine acridone acetate, which is an interferon inducer. Interferons are the most important system of innate immunity, which has antiviral and immunomodulatory effects, and can protect the body from infection with a virus, and in case of infection, fight the causative agent of the disease. The planned clinical trial of the efficacy and safety of the drug CYCLOFERON in the dosage form of a tablet will study its ability to prevent influenza and other respiratory viral infections in adults who have already had close contact with patients with manifest disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 65 years inclusive.
2. Written informed consent.
3. Co-living with persons who has developed influenza or other acute respiratory viral infection, diagnosed no more than 3 days ago.
4. No signs of acute respiratory viral infection, influenza or COVID-19 at the time of inclusion in the study.
5. For women with preserved reproductive potential - a negative pregnancy test and consent to use approved methods of contraception during the entire period of participation in the study; for men - consent to use approved methods of contraception during the entire period of participation in the study and for 3 weeks after the end of the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to meglumine acridone acetate and/or any other component of the drug/placebo.
2. Lactose intolerance
3. Diseases of the digestive system in the acute stage (erosions, gastric and/or duodenal ulcers, gastritis and duodenitis).
4. History of allergic reactions.
5. Decompensated liver cirrhosis.
6. Diseases of the thyroid gland.
7. Congenital or acquired immunodeficiency.
8. Signs of acute respiratory viral infection, influenza or COVID-19 at the time of inclusion.
9. Positive result of a rapid test for the presence of SARS-CoV-2 at the time of screening.
10. Vaccination to prevent COVID-19 and/or influenza within 6 months before screening, planned vaccination during a clinical trial.
11. History of positive test result for HIV types 1 or 2.
12. Pregnancy or breastfeeding period (for women).
13. Alcoholism, drug addiction, substance and/or drug abuse in history and/or at the time of screening.
14. Participation in another clinical trial within 3 months before inclusion.
15. Subject is already receiving cycloferon.
16. Subject is receiving prohibited therapy or was receiving it within 30 days prior to screening.
17. Failure to observe the subject during the study period.
18. Other reasons that, in the opinion of the researcher, prevent the subject from participating in the study or create an unreasonable risk (for example, a history of autoimmune diseases, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Proportion of influenza/other acute respiratory viral infection in the study groups | 14 days
  the proportion of subjects with clinically manifest and laboratory confirmed influenza or other acute respiratory viral infection, developed within days 1-14 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana V Kharitonova, MD PhD, Study Director — STPF POLYSAN
Locations (2):
- Russia (2):
  - Research Center for Eco-safety, Ltd., Saint Petersburg
  - City Outpatient Clinic #117, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No